CLINICAL TRIAL: NCT04580407
Title: A Phase 2/3, Open-Label, Non-controlled Study to Evaluate the Efficacy and Safety of B-Domain Deleted Recombinant Porcine Factor VIII (rpFVIII, TAK-672), in the Treatment of Serious Bleeding Episode in Japanese Subjects With Acquired Hemophilia A (AHA)
Brief Title: Study of TAK-672 in Participants With Acquired Hemophilia A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-672-3001; U1111-1258-0779 (Other: WHO); jRCT2051200066 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Acquired Hemophilia A
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-672 (Experimental): TAK-672 was administered at an initial dose of 200 U/kg with IV infusion at a rate of 1-2 mL/min at Day 1. Subsequent doses were determined based on the post-infusion FVIII:C achieved after the most recent dose given, the target FVIII:C, and pFVIII inhibitor titer.
  Interventions: Biological: TAK-672

INTERVENTIONS:
Biological: TAK-672 — B-Domain Deleted Recombinant Porcine Factor VIII
  Other Names: rpFVIII, TAK-672, Obizur

SUMMARY:
The main aims of the study are to learn if TAK-672 can control bleeds in participants with acquired hemophilia A and if the participants have side effects from TAK-672. Acquired hemophilia A is when people's immune system attacks specific proteins, known as clotting factors, in their bodies. This is different from hemophilia A, which is a condition people are born with.

At the first visit, the study doctor will check who can take part. For those who can take part, participants will visit the clinic or hospital when they get their next bleed. They will receive TAK-672 slowly through a vein. This is called an infusion. They might need extra infusions of TAK-672 to control the bleed. After their bleed is controlled, participants will regularly visit the clinic for a check-up and to treat any further bleeds. This will happen until all participants have received their last dose of TAK-672 to control their 1st bleed. After this, all participants will visit the clinic 90 days later for a final check-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Japanese participants of >=18 years of age.
2. Participants who (or their legally authorized representatives) have provided his/her written informed consent form prior to any study-related procedures and study product administration.
3. Participants with a diagnosis of AHA based on clinical evaluation and supportive local laboratory testing as shown below:

   * Presentation with spontaneous bleeding without anatomical cause and without prior known bleeding disorder.
   * Prolonged activated partial thromboplastin time (aPTT) without explanation.
   * Abnormal aPTT cross mixing test consistent with FVIII inhibitors
   * Confirmation of a low FVIII:C.
   * Positive FVIII inhibitor (>=0.6 BU) as measured either in the local or central laboratory
4. Participants with a severe bleeding episode which the investigator finds necessary to treat and whose severe bleeding episode meets at least 1 of the following criteria:

   * Bleeds that pose a threat to a vital organ that could threaten life (e.g. intracranial bleed, or any site that could obstruct the airway).
   * Bleeds that pose a threat to a vital organ where life is not threatened but the organ function could be impaired (e.g., intraspinal bleed threatening the spinal cord and/or nerve conduction; a continual bleed into the kidney or bladder that could result in an obstructive uropathy, testicular bleed, bleed in and around the eye).
   * Bleeds requiring a blood transfusion to maintain the Hgb level at above-life or organ threatening levels (e.g. post-surgical, gastro-intestinal, retro-peritoneal, and thigh bleeds).
   * Intramuscular bleeds where muscle viability and/or neurovascular integrity is significantly compromised or at risk of being compromised.
   * Intra-articular bleeds impacting a major joint associated with severe pain, swelling and severe loss of joint mobility (reduced >70%) or where a bleed could result in joint destruction (e.g. in and around the femoral head).
5. Participants who are taking anti-thrombotics (including anti-platelet agents and anticoagulantswith confirmatory laboratory testing documenting specific FVIII inhibitor titer and with 3 half-lives of the agent have elapsed since the last dose.
6. Participants with expected life expectancies of at least 90 days prior to the onset of the hemorrhagic episode.
7. Participants of reproductive age who have agreed to use acceptable methods of contraception and if female, undergo pregnancy testing as part of the screening process.
8. Participant who are able to willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participants with an established reason for bleeding that is not correctable even with hemostatic therapy.
2. Participants presenting a bleeding episode that is assessed likely to resolve on its own, even if left untreated.
3. Participants with a known major sensitivity (anaphylactoid reactions) to therapeutic products of porcine or hamster origin; examples include therapeutics of porcine origin (e.g. previously marketed porcine FVIII, Hyate: C) and recombinant therapeutics prepared from hamster cells (e.g. Humira, Advate, and Enbrel).
4. Participants with the use of hemophilia medication: prior to the administration of TAK-672 under one of the following conditions: (1) use of "recombinant activated factor VII (rFVI)Ia " within 3 hours prior to TAK-672 administration (2) use of " activated prothrombin complex concentrate (aPCC)" within 6 hours prior to TAK-672 administration or (3) use of " plasma-derived FX/FVIIa complex concentrate (pd-FX/FVIIa) " within 8 hours prior to TAK-672 administration.
5. Participants with an anticipated need for treatment or device during the study that may interfere with the evaluation of the safety or efficacy of TAK-672, or whose safety or efficacy may be affected by TAK-672.
6. Participants who are currently pregnant or breastfeeding, or planning to become pregnant or father a child during the study
7. Participants who have participated in another clinical study and has been exposed to an investigational product or device within 30 days prior to the study enrollment.
8. Participants who are scheduled to participate in another non-observational (interventional) clinical study involving an investigational product or device during the course of the study.
9. Participants who are unable to or unwilling to comply with the study design, protocol requirements, and/or the follow-up procedures.
10. Participants whose majority of age are under legal protection.
11. Participants who are an immediate family member, study site employee, or are in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g. spouse, parent, child, sibling) or may consent under duress.
12. Participants who are judged by the investigator as being ineligible for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- Japan (9):
  - Gunma University Hospital, Maebashi, Gunma
  - Nagoya University Hospital, Aichi, Nagoya
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Uonuma Kikan Hospital, Minamiuonuma, Niigata
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Saiseikai Central Hospital, Mita, Tokyo
  - Chiba University Hospital, Chiba
  - Fukushima Medical University Hospital, Fukushima
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f9464b2296beb001e63bf9f

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in Japan from 09 April 2021 to 29 November 2022.
Pre-assignment Details: A total of 5 participants with Acquired Hemophilia A (AHA) were enrolled in this study to receive TAK-672 at an initial dose of 200 units per kilogram (U/kg).
Groups:
- TAK-672: TAK-672 was administered at an initial dose of 200 U/kg with intravenous (IV) infusion at a rate of 1-2 milliliters per minute (mL/min) at Day 1. Subsequent doses were determined based on the post-infusion factor VIII activity (FVIII:C) achieved after the most recent dose given, the target FVIII:C, and pFVIII inhibitor titer.
Period: Overall Study
Arm/Group | TAK-672
Started | 5
Completed | 4
Not Completed | 1
Not completed — Judged to be Required to Receive Prophylactic Treatment with Emicizumab | 1

BASELINE CHARACTERISTICS:
Population: Full analysis Set (FAS) included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Arm/Group | TAK-672
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 154.1 (12.71)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 53.42 (7.529)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Severe Bleeding Episodes Who Demonstrated Response to TAK-672 Therapy at 24 Hours After the Initiation of Treatment
Description: Percentage of severe bleeding episodes with demonstrated response to TAK-672 therapy at 24 hours after the initiation of treatment was assessed by using a well-defined 4-point ordinal scale - A 'positive response' was defined as 'effective' (bleeding stopped with clinical control and FVIII:C levels of 50% or higher ) or 'partially effective' (bleeding reduced with clinical stabilization and FVIII:C levels of 20% or higher) control of bleeding, as determined by the investigator using a 4-point rating scale (effective - partially effective - poorly effective - not effective). 'Poorly effective' was defined as 'bleeding slightly reduced or unchanged and FVIII:C levels of less than 50%'. 'Not effective' was defined as 'bleeding worsening and FVIII:C levels of less than 20%'.
Time Frame: 24 hours after the initial dose of TAK-672
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
percentage of participants | 100 [47.818 to 100.000]

2. Secondary Outcome: Percentage of Participants With Severe Bleeding Episodes Successfully Controlled With TAK-672 Therapy, as Assessed by the Investigator
Description: If the status assessed by the investigator at the end of study treatment of initial treatment period was "successfully controlled", the participant's initial severe bleeding episode was considered as successfully controlled.
Time Frame: From first dose of study drug up to 90 days after the last dose of study drug or until discontinued (Up to 95 days as a maximum)
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
percentage of participants | 100 [47.818 to 100.000]

3. Secondary Outcome: Percentage of Participants With Bleeding Episodes Responsive to TAK-672 Therapy at Designated Assessment Time Points After the Initiation of Therapy, as Assessed by the Investigator
Description: A 'positive response' was defined as 'effective' (bleeding stopped with clinical control and FVIII:C levels of 50% or higher ) or 'partially effective' (bleeding reduced with clinical stabilization and FVIII:C levels of 20% or higher) control of bleeding, as determined by the investigator using a 4-point rating scale (effective - partially effective - poorly effective - not effective). 'Poorly effective' was defined as 'bleeding slightly reduced or unchanged and FVIII:C levels of less than 50%'. 'Not effective' was defined as 'bleeding worsening and FVIII:C levels of less than 20%'. Data is reported only for the timepoints having at least one participant available for analysis.
Time Frame: At 0.5, 8, 16, 24, 48, 60, 96, and 120 hours post dose and at 1, 14, 28, 42, 56, 70, and 90 day follow-up
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses. Number of participants analyzed are the number of participants available for analysis at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
percentage of participants
  Initial Treatment Period at 0.5 Hours | 80.0 [28.358 to 99.495]
  Initial Treatment Period at 8 Hours | 100 [47.818 to 100.000]
  Initial Treatment Period at 16 Hours: number analyzed (Participants) | 4
  Initial Treatment Period at 16 Hours | 100 [39.764 to 100.000]
  Initial Treatment Period at 24 Hours | 100 [47.818 to 100.000]
  Initial Treatment Period at 48 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 48 Hours | 100 [2.500 to 100.000]
  Initial Treatment Period at 60 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 60 Hours | 100 [2.500 to 100.000]
  Initial Treatment Period at 96 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 96 Hours | 100 [2.500 to 100.000]
  Initial Treatment Period at 120 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 120 Hours | 100 [2.500 to 100.000]
  Initial Treatment Period Follow-up at 24 Hours on Day 1 | 100 [47.818 to 100.000]
  Initial Treatment Period Follow-up at 14 Days | 100 [47.818 to 100.000]
  Initial Treatment Period Follow-up at 28 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 28 Days | 100 [39.764 to 100.000]
  Initial Treatment Period Follow-up at 42 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 42 Days | 100 [39.764 to 100.000]
  Initial Treatment Period Follow-up at 56 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 56 Days | 100 [39.764 to 100.000]
  Initial Treatment Period Follow-up at 70 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 70 Days | 100 [39.764 to 100.000]
  Initial Treatment Period Follow-up at 90 Days (End of Study): number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 90 Days (End of Study) | 100 [39.764 to 100.000]

4. Secondary Outcome: Frequency of Infusions Per Participant of TAK-672 Required to Successfully Control Qualifying Bleeding Episodes
Description: 'Frequency of infusions ' was calculated as the 'average number of infusions per day'. 'Qualifying bleeding episode' was defined as the 'initial, severe bleeding episode'.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: infusions per participant
Arm/Group | TAK-672
Number analyzed (Participants) | 5
infusions per participant | 1.8 (1.12)

5. Secondary Outcome: Total Dose of Infusions Per Participant of TAK-672 Required to Successfully Control Qualifying Bleeding Episodes
Description: 'Qualifying bleeding episode' was defined as the 'initial, severe bleeding episode'. Total dose of infusions is sum of doses from start of treatment with TAK-672 for qualifying bleeding episodes until completion of the management of the bleeding.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: dose per participant
Arm/Group | TAK-672
Number analyzed (Participants) | 5
dose per participant | 38640.0 (28442.45)

6. Secondary Outcome: Total Number of Infusions Per Participant of TAK-672 Required to Successfully Control Qualifying Bleeding Episodes
Description: 'Qualifying bleeding episode' was defined as the 'initial, severe bleeding episode'. If the status assessed by the investigator at the end of study treatment of initial treatment period was "successfully controlled", the participant's initial severe bleeding episode was considered as successfully controlled.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: infusions per participant
Arm/Group | TAK-672
Number analyzed (Participants) | 5
infusions per participant | 2.6 (0.89)

7. Secondary Outcome: Percentage of Participants With Response to TAK-672 Therapy at Specified Time Points and Eventual Control of Severe Bleeding Episodes
Description: Percentage of participants with response to TAK-672 therapy at specified time points and eventual control of severe bleeding episodes was assessed to determine the correlation between response to TAK-672 therapy and eventual control of severe bleeding episodes. A 'positive response' was defined as 'effective' (bleeding stopped with clinical control and FVIII:C levels of 50% or higher) or 'partially effective' (bleeding reduced with clinical stabilization and FVIII:C levels of 20% or higher) control of bleeding, as determined by the investigator using a 4-point rating scale (effective - partially effective - poorly effective - not effective). 'Poorly effective' was defined as 'bleeding slightly reduced or unchanged and FVIII:C levels of less than 50%'. 'Not effective' was defined as 'bleeding worsening and FVIII:C levels of less than 20%'. Data is reported only for the timepoints having at least one participant available for analysis.
Time Frame: At 0.5, 8, 16, 24, 48, 60, 96,120, and 144 hours post dose and at 1, 14, 28, 42, 56, 70, and 90 day follow-up
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
percentage of participants
  Initial Treatment Period at 0.5 Hours | 80.0
  Initial Treatment Period at 8 Hours | 100
  Initial Treatment Period at 16 Hours: number analyzed (Participants) | 4
  Initial Treatment Period at 16 Hours | 100
  Initial Treatment Period at 24 Hours | 100
  Initial Treatment Period at 48 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 48 Hours | 100
  Initial Treatment Period at 60 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 60 Hours | 100
  Initial Treatment Period at 96 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 96 Hours | 100
  Initial Treatment Period at 120 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 120 Hours | 100
  Initial Treatment Period at 144 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 144 Hours | 100
  Initial Treatment Period Follow-up at 24 Hours on Day 1 | 100
  Initial Treatment Period Follow-up at 14 Days | 100
  Initial Treatment Period Follow-up at 28 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 28 Days | 100
  Initial Treatment Period Follow-up at 42 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 42 Days | 100
  Initial Treatment Period Follow-up at 56 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 56 Days | 100
  Initial Treatment Period Follow-up at 70 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 70 Days | 100
  Initial Treatment Period Follow-up at 90 days (End of Study): number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 90 days (End of Study) | 100

8. Secondary Outcome: Mean Value of Pre-infusion Anti-TAK-672 Antibody Titers in Participants With Successful Control of the Bleeding Episode
Description: Mean value of pre-infusion anti-TAK-672 antibody titers (unit: Bethesda unit per milliliters [BU/mL]) in participants with successful control of the bleeding episode was reported as a result of correlation among the pre-infusion pFVIII inhibitor titers and the eventual control of the bleeding episode in this outcome measure.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: Bethesda unit per milliliters (BU/mL)
Arm/Group | TAK-672
Number analyzed (Participants) | 5
Bethesda unit per milliliters (BU/mL) | 3.78 (4.784)

9. Secondary Outcome: Mean Value of Total Dose Per Participant in Participants With Successful Control of the Bleeding Episode
Description: Mean value of total dose per participant for initial treatment period (unit: units/kg per participant) in participants with successful control of the bleeding episode was reported as a results of correlation among the total dose per participant of TAK-672 and the eventual control of the bleeding episode in this outcome measure.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: units/kg per participant
Arm/Group | TAK-672
Number analyzed (Participants) | 5
units/kg per participant | 38640.0 (28442.45)

10. Secondary Outcome: Number of Participants With Positive Response at 24 Hours After the Initiation of Treatment in Participants With Successful Control of the Bleeding Episode
Description: Number of participants with positive response at 24 hours after the initiation of treatment in participants with successful control of the bleeding episode was reported as a results of correlation among the response at 24 hours and the eventual control of the bleeding episode. A 'positive response' was defined as 'effective'(bleeding stopped with clinical control and FVIII:C levels of 50%or higher) or 'partially effective'(bleeding reduced with clinical stabilization and FVIII:C levels of 20%or higher) control of bleeding, as determined by investigator using 4-point rating scale (effective-partially effective-poorly effective-not effective).
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
Participants | 5

11. Secondary Outcome: Anti-hFVIII Inhibitor Titers
Description: Data is reported only for the timepoints having at least one participant available for analysis.
Time Frame: Baseline, 72 hours postdose, and at 14, 28, 42, 56, 70, and 90 days follow-up
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses. Number analyzed is the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: BU/mL
Arm/Group | TAK-672
Number analyzed (Participants) | 5
BU/mL
  Initial Treatment Period Baseline | 57.6 (55.24)
  Initial Treatment Period at 72 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 72 Hours | 60.0 (NA) — Standard Deviation (SD) was not estimable for 1 participant.
  Initial Treatment Period Follow-up at 14 Days | 35.0 (65.51)
  Initial Treatment Period Follow-up at 28 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 28 Days | 27.3 (51.84)
  Initial Treatment Period Follow-up at 42 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 42 Days | 44.0 (88.00)
  Initial Treatment Period Follow-up at 56 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 56 Days | 46.3 (92.50)
  Initial Treatment Period Follow-up at 70 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 70 Days | 53.8 (107.50)
  Initial Treatment Period Follow-up at 90 Days (End of Study): number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 90 Days (End of Study) | 52.0 (104.00)

12. Secondary Outcome: Anti-pFVIII Inhibitor Titer
Description: Data is reported only for the timepoints having at least one participant available for analysis.
Time Frame: Baseline, 72 hours postdose, and at 14, 28, 42, 56, 70, and 90 days follow-up
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: BU/mL
Arm/Group | TAK-672
Number analyzed (Participants) | 5
BU/mL
  Initial Treatment Period at Baseline | 3.78 (4.784)
  Initial Treatment Period at 72 Hours: number analyzed (Participants) | 1
  Initial Treatment Period at 72 Hours | 0.00 (NA) — SD was not estimable for 1 participant.
  Initial Treatment Period Follow-up at 14 Days | 1.34 (2.475)
  Initial Treatment Period Follow-up at 28 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 28 Days | 1.18 (2.350)
  Initial Treatment Period Follow-up at 42 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 42 Days | 2.23 (4.450)
  Initial Treatment Period Follow-up at 56 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 56 Days | 3.33 (6.650)
  Initial Treatment Period Follow-up at 70 Days: number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 70 Days | 3.68 (7.350)
  Initial Treatment Period Follow-up at 90 Days (End of Study): number analyzed (Participants) | 4
  Initial Treatment Period Follow-up at 90 Days (End of Study) | 3.13 (6.250)

13. Secondary Outcome: Terminal Half-life (t1/2) for TAK-672
Time Frame: Pre-dose and at multiple time points post-dose (up to 24 hours) after over 48 hours from the last treatment with TAK-672
Population: PK evaluation was planned however, no PK sample was collected in this study due to none of the participants gave consent for the same.
Arm/Group | TAK-672
Number analyzed (Participants) | 0

14. Secondary Outcome: Clearance (CL) for TAK-672
Time Frame: as for outcome 13
Population: as for outcome 13
Arm/Group | TAK-672
Number analyzed (Participants) | 0

15. Secondary Outcome: Volume of Distribution (Vd) for TAK-672
Time Frame: as for outcome 13
Population: as for outcome 13
Arm/Group | TAK-672
Number analyzed (Participants) | 0

16. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) for TAK-672
Time Frame: Pre-dose and at multiple time points post-dose (up to 24 hours) after over 48 hours from the last treatment with the initial dose of TAK-672
Population: as for outcome 13
Arm/Group | TAK-672
Number analyzed (Participants) | 0

17. Secondary Outcome: Maximum Drug Concentration (Cmax) Per Dose (Cmax/Dose) for TAK-672
Time Frame: as for outcome 13
Population: as for outcome 13
Arm/Group | TAK-672
Number analyzed (Participants) | 0

18. Secondary Outcome: Duration Period From Initial Dose of TAK-672 Until Completion of Hemostasis Control
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Median (Full Range); unit: days
Arm/Group | TAK-672
Number analyzed (Participants) | 5
days | 1.0 [1 to 5]

19. Secondary Outcome: Total Dose Per Participant From Initial Dose of TAK-672 Until Completion of Hemostasis Control
Description: Total dose is sum of doses from start of treatment with TAK-672 until completion of hemostasis control.
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: dose per participant
Arm/Group | TAK-672
Number analyzed (Participants) | 5
dose per participant | 38640.0 (28442.45)

20. Secondary Outcome: Number of Participants With New Qualified Severe Bleeding Episodes
Time Frame: as for outcome 2
Population: FAS included all participants who had received at least 1 dose of the TAK-672 and was used for the efficacy analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-672
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 90 days after the last dose of study drug or until discontinued (Up to 95 days as a maximum)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-672
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-672 (N=5)
Central hypothyroidism (Endocrine disorders) | 1
Cryoglobulinaemia (Vascular disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-672 (N=5)
Anal fissure (Gastrointestinal disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood urine present (Investigations) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Delirium (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vessel puncture site haemorrhage (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04580407/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04580407/SAP_001.pdf